CLINICAL TRIAL: NCT04403100
Title: Hydroxychloroquine and Lopinavir/ Ritonavir for Hospitalization and Mortality Reduction in Patients With COVID-19 and Mild Disease Symptoms: "The Hope Coalition"
Brief Title: Hydroxychloroquine and Lopinavir/ Ritonavir to Improve the Health of People With COVID-19: "The Hope Coalition - 1"
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardresearch (Other)
Collaborators: Cardresearch - Cardiologia Assistencial e de Pesquisa LTDA (Unknown); Cytel Inc. (Industry)
Responsible Party: Principal Investigator, Gilmar Reis, Director - Outpatient Research Clinic, Cardresearch
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID19_AMB_Brasil
Record Dates: First submitted 2020-05-23; First posted 2020-05-27 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: COVID-19; Coronavirus Infection; Virus Disease; Acute Respiratory Infection; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Virus Diseases; Severe Acute Respiratory Syndrome | interventions — Hydroxychloroquine; Lopinavir; Ritonavir

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to one of four treatment arms in a 1:1:1:1 ratio:
  1. Lopinavir / Ritonavir
  2. Hydroxychloroquine
  3. Lopinavir / Ritonavir + Hydroxychloroquine
  4. Placebo.
  We will use a centralized random allocation schedule, generated by computer and implemented using an online remote access system. Randomization will be stratified by participating basic health unit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational medical product will be packaged in similar bottles by a third party who will keep the allocation confidential until the end of the study. The bottles will be sealed and identified as "Research Product A, B and C" and with different colored labels. They will be randomly allocated among the participants. The research subjects, medical assistance, administrative and health staff will not have access to the contents of the bottles. The Arm Lopinavir/ ritonavir plus hydroxychloroquine will receive two of such bottles.
  At the end of the study, after the statistical analysis and DMSB meeting, it will then be requested from third party documentation on content of each bottle and then have arms identified.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hydroxychloroquine Sulfate (Active Comparator): Hydroxychloroquine 400 mg. Loading oral dose of 800 mg followed by orally dose of 400 mg/ day for the following 10 days
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets
- Lopinavir/ Ritonavir (Active Comparator): Lopinavir Ritonavir 200/ 50 mg Loading oral dose of 800/ 200 mg twice a day on day 1 followed by 400/100 mg orally twice a day for the following 9 days
  Interventions: Drug: Lopinavir/ Ritonavir Oral Tablet
- Hydroxychloroquine plus Lopinavir/ Ritonavir (Active Comparator): Hydroxychloroquine 400 mg. Loading oral dose of 800 mg followed by orally dose of 400 mg/ day for the following 10 days
  Plus
  Lopinavir Ritonavir 200/ 50 mg Loading oral dose of 800/ 200 mg twice a day on day 1 followed by 400/100 mg orally twice a day for the following 9 days
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets plus Lopinavir/ Ritonavir Oral Tablets
- Placebo (Placebo Comparator): Placebo
  Twice a day from day 1 through day 10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate Tablets — Tablets of 400 mg: Loading dose of 02 tablets followed by one tablet of 400 mg orally on the following 09 days
  Arms: Hydroxychloroquine Sulfate
Drug: Lopinavir/ Ritonavir Oral Tablet — tablets of 200/ 50 mg; Loading dose of 04 tablets twice a day on day 1 followed by two tablets twice a day on the following 09 days
  Arms: Lopinavir/ Ritonavir
Drug: Hydroxychloroquine Sulfate Tablets plus Lopinavir/ Ritonavir Oral Tablets — Hydroxychloroquine Oral Tablet 400 mg: Loading dose of 02 tablets followed by one tablet of 400 mg orally on the following 09 days
  plus
  Lopinavir/ Ritonavir Oral Tablet of 200/ 50 mg: Loading dose of 04 tablets twice a day on day 1 followed by two tablets twice a day on the following 09 days
  Arms: Hydroxychloroquine plus Lopinavir/ Ritonavir
Drug: Placebo — Placebo tablets - 01 tablet twice daily from day 01 through day 10.
  Arms: Placebo

SUMMARY:
The COVID-19 pandemic has been characterized by high morbidity and mortality, especially in certain subgroups of patients. To date, no treatment has been shown to be effective in controlling this disease in hospitalized patients with moderate and / or severe cases of this disease. Hydroxychloroquine and lopinavir / ritonavir have been shown to inhibit SARS-CoV viral replication in experimental severe acute respiratory symptoms models and have similar activity against SARS-CoV2. Although widely used in studies of critically ill patients, to date, no study has demonstrated its role on the treatment of high-risk, newly diagnosed patients with COVID-19 and mild symptoms.

DETAILED DESCRIPTION:
In December 2019 a series of viral pneumonia cases were reported in the city of Wuhan, China. A new subtype of coronavirus has been identified as the causative agent of this condition. On February 11, 43,103 cases had already been described and on this day the World Health Organization (WHO) named this disease as COVID-19. With. The disease had spread out to several countries on different continents and on March 11, WHO declared a state of worldwide pandemic. Today (April 25, 2020) there are 2,719,897 cases and 187,705 deaths documented, with a global case-fatality ratio of 6.9%.

To date, no treatment has been identified as effective in combating this disease which has been identified as with high mortality, therefore there are no specific therapeutic options. So far, efforts have been focused on the treatment of patients hospitalized with dyspnea and, although several promising drugs are being evaluated, none has demonstrated effectiveness in reducing morbidity and mortality at this stage of the disease, suggesting that perhaps the best time to use medications either before the onset of severe symptoms of respiratory distress.

Thus, we propose the use of two drugs which experimentally have shown activity against SARS-CoV2 and being used in severely ill patients with COVID-19. Our hypothesis is that perhaps using such drugs before onset of complications will allow better outcomes on this patient population.

ELIGIBILITY:
Inclusion Criteria:

Patients with RT-PCR diagnosis of COVID-19 or a clinical condition compatible with COVID-19 and respiratory symptoms, presenting:

A. Persistent dry cough associated with axillary temperature > 37.7 Celsius;

OR

B. Recent onset of Flu-like Respiratory Symptoms associated with dry cough

OR

C. Tomographic image compatible with COVID 19 infection;

2. Men and women aged > 50 years OR: Patients over 18 years of age with at least one of the following criteria

* Diabetes requiring oral medication or insulin.
* Arterial hypertension requiring at least 01 oral medication for treatment
* Known cardiovascular diseases (CHF of any etiology, documented Coronary Artery Disease, Clinically overt heart disease)
* Symptomatic chronic lung disease and/ or medically controlled
* Patients with a history of transplantation
* Patient with stage IV chronic kidney disease or on dialysis.
* Patients on current Immunosuppression and/or using corticosteroid therapy (equivalent to at least 10 mg of oral prednisone per day)
* Willingness to comply with study related procedures

  3. Ability to provide informed consent before any protocol-related procedures.

Exclusion Criteria:

1. RT-PCR exam for COVID-19 negative during the screening visit.
2. Patients with an acute respiratory condition compatible with COVID-19 being hospitalized;
3. Patients with an acute respiratory condition and with moderate to high probability of not being a COVID infection 19;
4. Dyspnea secondary to other acute and chronic respiratory causes or infections (eg, decompensated Chronic Obstructive Pulmonary Disease, acute bronchitis, pneumonia, primary pulmonary arterial hypertension);
5. Severe respiratory clinical condition, presenting at least ONE of the criteria below:

   1. Respiratory Rate> 28 / min;
   2. Arterial Oxygen Saturation < 92% with nasal oxygen therapy at 10 l/ min;
   3. PaO2 / FIO2 <300 mmHg

4. History of Cardiac Arrhythmia or Long QT Syndrome; 5. Use of Medications that are known to prolong QTc: Citalopram, Venlafaxine, Bupropion and with no possibility of suspension during the period of investigational medical product administration. 6. Inability to take oral medications; 7. Patients on continuous use of Amiodarone and / or PGE5 Inhibitors (Ex .: Sildenafil and similar). 8. Use of Digoxin, Cyclosporine, Cimetidine, Tamoxifen. 9. Use of anticonvulsants, antifungals, immunosuppressants other than corticotherapy. 10. Use of Hydroxychloroquine for other indications 11. Use of chemoprophylaxis for malaria. 12. Psoriasis in a form other than cutaneous 13. Porphyria 14. Use of protease inhibitors, ritonavir or Cobicistat 15. Clinical history of Liver Cirrhosis or Child-Pugh C classification; 16. Patients with a history of degenerative retinal diseases (patients with retinal diseases due to diabetes and hypertension can participate in the research); 17. Patient with a clinically relevant history of hearing loss; 18. Patients with known severe degenerative neurological diseases and / or severe mental illness; 19. Inability of the patient or representative to give consent or adhere to the procedures proposed in the protocol; 20. Known hypersensitivity and / or intolerance to Hydroxychloroquine. 21. Hypersensitivity and / or intolerance Lopinavir / Ritonavir

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1968 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who were hospitalized for progression of COVID-19 disease | Measuring during 28-day period since randomization (Intention to treat analysis)
  Hospitalization is defined as at least 24 hours of acute care in a hospital or similar acute care facility (emergency settings, temporary emergency facilities created for acute care of COVID-19 pandemic)
Proportion of participants who died due to COVID-19 progression and/ or complications | Measuring during 28-day period since randomization (Intention to treat analysis)

SECONDARY OUTCOMES:
Proportion of participants with viral load change on 03, 07, 10 and 14 after randomization | Measuring during 14-day period since randomization
  Viral load change on 03, 07, 10 and 14 after randomization (200 patients per arm)
Time to clinical improvement | Measuring during 28-day period since randomization
  Proportion of participants with clinical improvement, defined as normalization of temperature, Respiratory rate, SaO2, and cough relief (> 50% compared to baseline measured on a visual analog scale) in the last 72 hours.
Time to clinical failure | Measuring during 28-day period since randomization
  Proportion of participants with clinical improvement, defined as as time to need for hospitalization due to dyspnea, death, need for mechanical ventilation, shock and need for vasoactive amines;
Hospitalization for any cause | Measuring during 28-day period since randomization
  Proportion of participants with hospitalization for any cause
Proportion of participants who died due to pulmonary complications | Measuring during 28-day period since randomization
Proportion of participants who died due to cardiovascular complications | Measuring during 28-day period since randomization
Proportion of participants who presented with adverse events | Measuring during 28-day period since randomization
  Evaluation of adverse events evaluated as associated to any of study arms
Time to improvement on respiratory scale symptoms | Measuring during 28-day period since randomization
  Proportion of participants who presented sustained improvement on respiratory scale defined as at least 48 hours of improvement.
proportion of non-adherent participants to any of study drugs | Measuring during 10-day period since randomization

CONTACTS AND LOCATIONS:
Overall Officials: Gilmar Reis, MD, PhD, Principal Investigator — Cardresearch - Cardiologia Assistencial e de Pesquisa LTDA
Locations (4):
- Brazil (4):
  - CARDRESEARCH - Cardiologia Assistencial e de Pesquisa, Belo Horizonte, Minas Gerais
  - Pontificia Universidade Catolica de Minas Gerais, Belo Horizonte, Minas Gerais
  - Fundo Municipal de Saúde de Betim, Betim, Minas Gerais
  - Universidade Federal de Ouro Preto, Ouro Preto, Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reis G, Moreira Silva EADS, Medeiros Silva DC, Thabane L, Singh G, Park JJH, Forrest JI, Harari O, Quirino Dos Santos CV, Guimaraes de Almeida APF, Figueiredo Neto AD, Savassi LCM, Milagres AC, Teixeira MM, Simplicio MIC, Ribeiro LB, Oliveira R, Mills EJ; TOGETHER Investigators. Effect of Early Treatment With Hydroxychloroquine or Lopinavir and Ritonavir on Risk of Hospitalization Among Patients With COVID-19: The TOGETHER Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e216468. doi: 10.1001/jamanetworkopen.2021.6468. PMID 33885775